CLINICAL TRIAL: NCT01667380
Title: Non-interventional Study on the Use of Mircera in the Treatment of Chronic Renal Anemia in Patients With Chronic Kidney Disease Stages III-IV Not on Dialysis and in Patients on Stage V on Hemodialysis
Brief Title: An Observational Study of Mircera in Patients With Chronic Renal Anemia on Dialysis (CKD Stage V) or Not on Dialysis (CKD Stage III-IV)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25617
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the use and efficacy of Mircera (methoxy polyethylene glycol-epoetin beta) in anemia patients with chronic kidney disease (CKD) stage III-IV not on dialysis or CKD stage V on dialysis. Patients will be followed during 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with chronic renal anemia with stage III-IV CKD not on dialysis and who are, in the opinion of the treating physician, not expected at baseline to require dialysis within 12 months
* Patients with chronic renal anemia with stage V CKD on dialysis
* No contraindication to ESA treatment

Exclusion Criteria:

* Uncontrolled hypertension
* Hypersensitivity to the active substance or any other of the excipients of Mircera and other ESAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anemia patients with chronic kidney disease (CKD) stage III-IV not on dialysis or CKD stage V on dialysis
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Dosage/schedule of Mircera treatment in clinical practice | approximately 3 years

SECONDARY OUTCOMES:
Proportion of patients with mean Hb level 10-12 g/dL 10 to 12 months after initiation of treatment | approximately 3 years
Change in Hb levels | from baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Podgorica, Montenegro